CLINICAL TRIAL: NCT01844076
Title: Quinacrine-Capecitabine Combinatorial Therapy for Advanced Stage Colorectal Adenocarcinoma:A Phase I/II Investigator-Initiated Clinical Trial
Brief Title: Quinacrine-Capecitabine Combinatorial Therapy for Advanced Stage Colorectal Adenocarcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The single Quinacrine manufacture facility in the US was shut down by the FDA
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GI-078
Record Dates: First submitted 2013-03-04; First posted 2013-05-01 (Estimated); Results first posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Colorectal Adenocarcinoma
Keywords: advanced stage colorectal adenocarcinoma
MeSH Terms: interventions — Quinacrine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase I Level -2 (Experimental): Phase I (Quinacrine and Capecitabine): The Phase I portion of the study will aim to determine the tolerability of both agents in combinations when used at established clinical doses. This portion of the study will more closely resemble a pilot study or feasibility study rather than a dose escalation.
  Each group will have 1 to 6 patients enrolled in it. If the patients in a lower group do not have any significant side effects the next patient will start at the next group dose.
  Group 1: capecitabine at a dose of 1000 mg/m^2 twice per day (days 1-14), and quinacrine at a dose of 100 mg once per day (days 1-21) for a 21 day cycle
  Interventions: Drug: Quinacrine and Capecitabine
- Phase I Level -1 (Experimental): Phase I (Quinacrine and Capecitabine): The Phase I portion of the study will aim to determine the tolerability of both agents in combinations when used at established clinical doses. This portion of the study will more closely resemble a pilot study or feasibility study rather than a dose escalation.
  Each group will have 1 to 6 patients enrolled in it. If the patients in a lower group do not have any significant side effects the next patient will start at the next group dose.
  Group 1: capecitabine at a dose of 1000 mg/m^2 twice per day (days 1-14), and quinacrine at a dose of 100 mg twice per day (days 1-21) for a 21 day cycle
  Interventions: Drug: Quinacrine and Capecitabine
- Phase I Level 0 (Experimental): Group 3: capecitabine at a dose of 1000 mg/m^2 twice per day (days 1-14), quinacrine at a dose of 200 mg twice a day (days 1-21) for a 21 day cycle
  Interventions: Drug: Quinacrine and Capecitabine
- Phase II (Experimental): Phase II will use the treatment outlined in phase I, using the recommended phase II dose (RP2D) derived from Phase I.
  Patients will receive capecitabine at a dose of 1000 mg/m^2 twice per day (days 1-14), quinacrine at a dose of 100 mg twice per day (days 1-21) for a 21 day cycle
  Interventions: Drug: Quinacrine and Capecitabine

INTERVENTIONS:
Drug: Quinacrine and Capecitabine — The Phase I portion of the study will aim to determine the tolerability of both agents in combinations when used at established clinical doses. This portion of the study will more closely resemble a pilot study or feasibility study rather than a dose escalation.
  Other Names: Quinacrine; Capecitabine

SUMMARY:
Establish the tolerability and safety of aimed dose of both quinacrine and capecitabine in combination to treat patients with advanced colorectal adenocarcinoma.

DETAILED DESCRIPTION:
Because of the well published safety profiles of both quinacrine and capecitabine, the Phase I portion of our study will aim to determine the tolerability of both agents in combinations when used at established clinical doses. This portion of the study will more closely resemble a pilot study or feasibility study rather than a dose escalation Phase I trial. The objective is to determine toxicities and adverse reactions, not a maximally tolerated dose. The investigators hypothesize that there will be no toxic interactions at the pharmacokinetic or pharmacodynamic level, and want to know the feasibility of using quinacrine and capecitabine at their respective recommended single agent doses. Because capecitabine is already regarded as standard treatment for colorectal cancer, the investigators will begin the study with a full dose of capecitabine combined with a slightly lower dose of quinacrine. If the safety-interim analysis does not detect an excess of toxicity, then subsequent patients will be enrolled using the full dose of both drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients much have histologically confirmed adenocarcinoma of the colon or rectum.
* Patients must have measurable recurrence or metastases in the liver and/or lungs.
* Patients must have prior chemotherapy for advanced colorectal cancer and have previously received both an oxaliplatin and an irinotecan based regimen.
* Age > 18 years.
* Life expectancy greater than 4 weeks.
* ECOG performance status <3.
* Patients must have normal organ and marrow function.
* Patients must be able to swallow capsules.
* Patients must be able to understand and willing to sign a written informed consent document.
* Patients are included regardless of KRAS/BRAF status.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients may not be receiving any other investigational agent.
* Patients with know brain metastases should be excluded from this clinical trial because they often develop progressive neurological dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to quinacrine, capecitabine or fluorouracil.
* The concomitant use of quinacrine and primaquine is contraindicated.
* Uncontrolled intercurrent illness including but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study.
* Patients with a baseline creatinine clearance of < 50 mL/min.
* Patients must be currently not treated with quinacrine or drugs related to quinacrine.
* Patients who require anti-arrhythmic treatment with amiodarone or any drug with a quinidine-like effect on the heart or who have history of a malignant ventricular arrhythmia unless they have a functioning automatic implantable cardio defibrillator implanted.
* Patients who have a history of noninfectious hepatitis or alcoholism.
* Patients with a lifetime history of porphyria or psoriasis because it can exacerbate these conditions.
* Patients with documented glucose-6-phosphate dehydrogenase deficiency.
* Patients with a lifetime history of seizure disorder.
* Patients with a lifetime history of dermatitis as an allergic/toxic reaction to any medication.
* Patients with know dihydropyrimidine dehydrogenase deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Crystal S. Denlinger, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Started study at new Institution

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Level -1: Group 2: capecitabine at a dose of 1000 mg/m^2 twice per day (days 1-14), quinacrine at a dose of 100 mg twice per day (days 1-21) for a 21 day cycle
- Phase II: Phase II will use the treatment outlined in phase I, using the RP2D derived from Phase I.
  Patients will receive capecitabine at a dose of 1000 mg/m^2 twice per day (days 1-14), quinacrine at a dose of 100 mg twice per day (days 1-21) for a 21 day cycle
Period: Overall Study
Arm/Group | Phase I Level -2 | Phase I Level -1 | Phase I Level 0 | Phase II
Started | 3 | 6 | 3 | 7
Completed | 1 | 6 | 3 | 7
Not Completed | 2 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Of the 19 patients enrolled in the study, two were not analyzed. One patient withdrew before receiving treatment, the other patient received no further treatment after a grade 3 toxicity at C1D1.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Level -2 | Phase I Level -1 | Phase I Level 0 | Phase II | Total
Number analyzed (Participants) | 1 | 6 | 3 | 7 | 17
Age, Continuous [Median (Full Range); unit: years] | 77 [77 to 77] | 56.5 [46 to 73] | 61 [54 to 66] | 61 [35 to 76] | 61 [35 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 1 | 1 | 6
  Male | 1 | 2 | 2 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 1 | 5 | 3 | 6 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 6 | 3 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Phase I - Number of Participants Who Experienced Dose Limiting Toxicities and Adverse Reactions
Description: Establish the tolerability of both agents in combination when used at established clinical doses. The objective is to determine toxicities and adverse reactions of patients in each group with different dose levels to find the maximum tolerated dose (MTD).
Time Frame: One year
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Level -2 | Phase I Level -1 | Phase I Level 0
Number analyzed (Participants) | 1 | 6 | 3
Participants | 0 | 0 | 3

2. Secondary Outcome: Phase II - Rate of Response
Description: Determine rate of response in patients receiving quinacrine in combination with capecitabine. Using Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) complete response (CR) is a disappearance of all target lesions, partial response (PR) is at least 30% decrease in the sum of diameters of target lesions, and overall response is the number of patients who experience a complete response or partial response.
Time Frame: 2-3 years
Population: Rate of response was analyzed for participants in phase II
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Level -2 | Phase I Level -1 | Phase I Level 0 | Phase II
Number analyzed (Participants) | 0 | 0 | 0 | 7
Participants | 0 | 0 | 0 | 1

3. Other Pre Specified Outcome: Phase II - Time to Progression (TTP)
Description: Determine time to progression from start of treatment in patients receiving quinacrine in combination with capecitabine. Using Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1), progression is defined as a 20% increase in sum of target lesions, with at least a 5 mm absolute increase.
Time Frame: 2-3 years
Population: TTP was analyzed for participants enrolled in phase II
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I Level -2 | Phase I Level -1 | Phase I Level 0 | Phase II
Number analyzed (Participants) | 0 | 0 | 0 | 7
months |  |  |  | 2.12 [1.85 to 4]

ADVERSE EVENTS:
Time Frame: 38 months
Arm/Group | Phase I Level -2 | Phase I Level -1 | Phase I Level 0 | Phase II
All-Cause Mortality (participants affected / at risk) | 1/1 | 5/6 | 3/3 | 6/7
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/6 | 2/3 | 2/7
Other Adverse Events (participants affected / at risk) | 1/1 | 6/6 | 3/3 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Level -2 (N=1) | Phase I Level -1 (N=6) | Phase I Level 0 (N=3) | Phase II (N=7)
Hospitalization (General disorders) | 0 | 0 | 1 | 0 — Dehydration, hyperkalemia, cough, generalized weakness
Hospitalization (General disorders) | 0 | 0 | 1 | 0 — Hepatic encephalopathy, melena, anemia
Hospitalization (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 — Hyponatremia, hyperbilirubinemia
Death (General disorders) | 0 | 0 | 1 | 0 — Hepatic encephalopathy, elevated ammonia level
Hospitalization (General disorders) | 0 | 1 | 0 | 0 — Abdominal pain, atrial fibrillation
Hospitalization (General disorders) | 0 | 1 | 0 | 0 — Pulmonary embolism, dyspnea, right leg dvt, acute kidney injury, right urethral obstruction
Hsopitalization (General disorders) | 0 | 1 | 0 | 0 — Nausea, vomiting, diarrhea, urinary tract infection, hydroureteronephrosis
Hospitalization (General disorders) | 0 | 0 | 0 | 1 — Nausea, vomiting, abdominal pain, bowel obstruction, parastomal hernia
Hospitalization (General disorders) | 0 | 0 | 0 | 1 — Deep vein thrombosis, acute kidney injury, edema in LLE
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Level -2 (N=1) | Phase I Level -1 (N=6) | Phase I Level 0 (N=3) | Phase II (N=7)
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2
Oral thrush (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 2 | 7
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 2 | 2
Hypertension (Vascular disorders) | 1 | 0 | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0 | 3 | 2
Hyperbilirubinemia (Investigations) | 1 | 1 | 2 | 0
Elevated AST (Investigations) | 1 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 1 | 1
Weight loss (Investigations) | 1 | 1 | 3 | 3
Burping (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 3 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 4 | 1 | 3 — Yellowing of skin
Urine discoloration (Renal and urinary disorders) | 0 | 1 | 0 | 0 — dark urine
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 4
Eye disorder - other (Eye disorders) | 0 | 1 | 0 | 0 — yellowing of eyes
Chills (General disorders) | 0 | 1 | 1 | 3
Nausea (Gastrointestinal disorders) | 0 | 4 | 3 | 3
Vomiting (Gastrointestinal disorders) | 0 | 2 | 2 | 4
Constipation (Gastrointestinal disorders) | 0 | 3 | 2 | 5
Polydipsia (General disorders) | 0 | 1 | 0 | 0
Mucositis (Gastrointestinal disorders) | 0 | 3 | 1 | 0
Edema (General disorders) | 0 | 4 | 1 | 1 — Limbs
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
ANC decreased (Investigations) | 0 | 1 | 1 | 0
ALT increased (Investigations) | 0 | 1 | 1 | 0
AST increased (Investigations) | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Peeling skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Increased ALP (Investigations) | 0 | 0 | 2 | 2
Pain - biliary tube (General disorders) | 0 | 0 | 1 | 0
Loss of consciousness (General disorders) | 0 | 0 | 1 | 0
Jaundice (General disorders) | 0 | 1 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Melena (General disorders) | 0 | 0 | 1 | 0
Weight gain (Investigations) | 0 | 0 | 1 | 0
Sweats (General disorders) | 0 | 0 | 1 | 3
Pulled muscle (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Numbness (General disorders) | 0 | 0 | 1 | 0 — Jaw
Dry eyes (Eye disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 — Hands
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1
Diziness (Nervous system disorders) | 0 | 1 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Burning sensation (General disorders) | 0 | 0 | 0 | 1
Small bowel obstruction (General disorders) | 0 | 0 | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 3
Deep vein thrombosis (General disorders) | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Edema (General disorders) | 0 | 0 | 1 | 0 — Trunk
Oral dysesthesia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nocturia (General disorders) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2
Lip swelling (General disorders) | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 1
Bilateral pulmonary embolism (Vascular disorders) | 0 | 1 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1
Cold sensitivity (Nervous system disorders) | 0 | 0 | 0 | 1
Dry heaving (Gastrointestinal disorders) | 0 | 1 | 1 | 0

LIMITATIONS AND CAVEATS:
Uncertain optimal time of peak plasma concentrations due to sample measurements at only 4 time points. Inaccurate half-life of Cmax due to lack of samples. Technical errors for lower-than-expected concentrations in participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/76/NCT01844076/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/76/NCT01844076/Prot_SAP_001.pdf